CLINICAL TRIAL: NCT04113187
Title: Study of the Efficacy of Propranolol for the Management of Epistaxis in Hereditary Hemorrhagic Telangiectasia Patients
Brief Title: Propranolol for Epistaxis in Hereditary Hemorrhagic Telangiectasia Patients
Acronym: EPERO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: AMRO-HHT-France - Association Maladie de Rendu-Osler (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX 2015/32
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Osler Weber Rendu Disease
Keywords: angiogenesis; epistaxis; propranolol
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol arm (Experimental)
  Interventions: Drug: Propranolol treatment
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol treatment — 40 mg twice a day (morning and evening), per os, during three months
  Arms: Propranolol arm
Drug: Placebo — per os, twice a day (morning and evening) during three months
  Arms: Placebo arm

SUMMARY:
Hereditary Hemorrhagic Telangiectasia (HHT) is a genetic disorder of angiogenesis associated with disabling epistaxis. Management of these nose bleedings requires more effective treatment. Propranolol, a beta-blocker, is a potentially useful therapeutic considering its anti-angiogenic properties. Our objective is to explore the efficacy of propranolol, three months after its introduction, on the cumulative duration of epistaxis in HHT patients.

DETAILED DESCRIPTION:
Hereditary Hemorrhagic Telangiectasia (HHT) is a rare systemic autosomal dominantly inherited disorder of angiogenesis. Its major feature is the occurrence in 90% of patients of spontaneous and recurrent epistaxis responsible for iron deficiency and chronic anemia. Various conservative and interventional treatments have been described for these conditions, but no optimal therapy exists. Inhibiting angiogenesis process is an interesting therapeutic option. Propranolol, a non-cardio-selective beta-blocker, could represent a new candidate for the therapy of HHT telangiectasia as it suppresses angiogenesis in vitro. This anti-angiogenic property is well-known in pediatric dermatology, since C. Léauté-Labrèze and al. have demonstrated a great improvement of infantile hemangioma undergoing propranolol treatment. At the University Hospital Center of Bordeaux, the investigators assessed in a preliminary study the efficacy of propranolol for HHT epistaxis. Nine of ten patients receiving propranolol for cardiologic or neurologic indications, retrospectively analyzed, significantly improved their Epistaxis Severity Score. Ten patients were then prospectively included and after 3 months of propranolol treatment, the median duration of epistaxis per month significantly decreased (p=0,007) as well as the number of epistaxis episodes per month (p=0,015).

To confirm these results, the investigators would like to study the efficacy of propranolol given per os at the dose of 40 mg twice a day for a three-months period, in comparison to a placebo. Throughout the study, patients will complete specific grids recording the number of epistaxis episodes per month and the cumulative duration of nose bleedings. A follow-up of 6 months will be done (4 visits after inclusion), recording clinical and biological data and monitoring the tolerance of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of HHT : 3 or more Curaçao criteria (spontaneous and recurrent epistaxis; multiple telangiectasia at characteristic sites; visceral lesions such as gastrointestinal telangiectasia or arteriovenous malformations; family history: a first degree relative with HHT according to these criteria ) or mutations of genes encoding for ALK1, ENG or SMAD4
* Patient suffering from recurrent epistaxis (more than a mean of 10 episodes/month) and/or with a cumulative mean duration per month more than 20 minutes, according to specific grids completed at least three months before inclusion.
* Patient insured under the French social security system
* Free and informed consent signed by investigator and patient

Exclusion Criteria:

* Pregnancy or breast-feeding
* Incomplete epistaxis grids in the month prior inclusion
* Current beta-blocker treatment
* Hypersensitivity to the active substance or excipient
* Patients with type I or type II diabetes, treated with insulin, sulphonylureas or meglitinides
* Patients with heart failure
* Patients with liver failure
* Patients with hepatic arteriovenous malformations responsible for high-output cardiac failure or severe hepatic dysfunction
* Patients with severe psoriasis (PASI>10)
* Contra-indication to beta-blocker treatment : asthma, chronic obstructive bronchopneumopathy, atrioventricular block of second or third degrees without pacemaker, Prinzmetal's angina, bradycardia < 50bpm, Raynaud's phenomenon, oblitering arteriopathy of the lower limbs, low blood pressure, non-treated pheochromocytoma
* Participation in another clinical therapeutic trial less than 3 months before inclusion
* Protected adult according to french law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Cumulative duration of epistaxis (in minutes) | 6 months after baseline (Day 0)

SECONDARY OUTCOMES:
Frequency of epistaxis (number of episodes) per month | At baseline (Day 0), 3 months and 6 months after baseline
Number of cutaneous telangiectasia on hands and face | At baseline (Day 0), 3 months and 6 months after baseline.
Levels of hemoglobin | At baseline (Day 0), 3 months and 6 months after baseline.
Levels of ferritin | At baseline (Day 0), 3 months and 6 months after baseline.
Number of red blood cells transfusions | At baseline (Day 0), 3 months and 6 months after baseline.
Short Form (SF) 36 Health Survey | At baseline (Day 0), 3 months and 6 months after baseline.
Number of adverse events | 3 months and 6 months after baseline (Day 0).
Measurement of blood pressure | At baseline (Day 0), 1 month, 3 months and 6 months after baseline.
Measurement of heart rate | At baseline (Day 0), 1 month, 3 months and 6 months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anne CONTIS, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de médecine interne, Bordeaux, France